CLINICAL TRIAL: NCT05704452
Title: Validity and Reliability of the Turkish Version of General Practitioner Assessment of Cognition
Brief Title: Validity and Reliability of the GPCOG -TR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: GPCOG Validity
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Dementia
Keywords: General Practitioners; Early diagnosis
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patient group: who diagnosed with dementia
- Control group: who diagnosed as healthy (don't have dementia)

SUMMARY:
The General Practitioner assessment of Cognition (GPCOG) was specifically developed as a brief cognitive screening tool to be used by general practitioners (GPs). It consists of a patient section testing cognition and an informant section asking historical questions. The aim of this study was to test the validity and reliability of the Turkish version of GPCOG-TR on Turkish older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age: least 55 years old
* Provide informed consent
* Diagnosed with dementia ( patient group)

Exclusion Criteria:

* Living in a nursing home
* Presence of psychiatric disorders requiring treatment
* Presence of other comorbidity interfering with cognitive performance such as severe chronic heart failure, chronic obstructive pulmonary disease, diabetes, anemia Impairment of auditory or visual perception
* Low education
* Known cognitive impairment (for control group only)
* Lack of a reliable informant.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: The participants of this study were members of the Neurology Department of Maltepe University Medical Faculty Hospital.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
The Clinical Dementia Rating score (CDR) | 1-2 hrs
  The scoring system from 0 to 3 ( 0 means healthy while 3 Severe dementia )
the General Practitioner Cognitive Assessment tool (GPCOG-TR) | 10 min
  Total score: 15
  * 9 for the patient part
  * 6 for the informant part ( The lower the score the more serious is the cognition is)

SECONDARY OUTCOMES:
The Mini-mental State Examination (MMSE) | 10 min
  Total score : 30
  Scores of 25-30 out of 30 are considered normal, 21-24 as mild, 10-20 as moderate and below 10 as severe impairment.
Alzheimer's Disease Assessment Scale-Cognitive scale (ADAS-Cog) | 30 min
  The total ADAS-Cog score ranges from 0-70 with higher scores suggesting greater impairment.
Geriatric Depression Scale (GDS) | 5 min
  Total score : 15
  0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)